CLINICAL TRIAL: NCT06239415
Title: PRospective Observational Study on PAtients With Symptomatic Peripheral Artery Disease on Rivaroxaban-acetylsalicylic Acid Combination Therapy (PRO-PAS)
Brief Title: PAtients With Symptomatic Peripheral Artery Disease on Rivaroxaban-acetylsalicylic Acid Combination Therapy (PRO-PAS)
Acronym: PRO-PAS
Status: Recruiting | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Società Italiana Cardiologia Ospedalità Accreditata (SICOA) (Unknown)
Responsible Party: Principal Investigator, Laura Adelaide Dalla Vecchia, Principal Investigator, Istituti Clinici Scientifici Maugeri SpA
Other Study IDs: 2605CE
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Peripheral Atherosclerotic Disease
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observation — Observation for 1 year of patients suffering from symptomatic peripheral atherosclerotic disease of the lower limb, with or without chronic ischemic heart disease, and indication for treatment with rivaroxaban 2.5 mg bid and acetylsalicylic acid 100 mg.

SUMMARY:
The observational, prospective, multicenter study enrolls patients experiencing symptomatic peripheral atherosclerotic disease in the lower limb, with or without chronic ischemic heart disease, and who have an indication for treatment with rivaroxaban 2.5 mg twice daily and ASA 100 mg. The study's objective is to assess adherence to the prescribed treatment after 3 months and 12 months from enrollment, as well as to monitor any adverse events that may occur during this period.

DETAILED DESCRIPTION:
Life expectancy in patients suffering from chronic peripheral obstructive arterial disease is significantly reduced compared to their non-arteriopathic peers. Mortality 15 years after diagnosis of ACOP is approximately 70%. Literature studies showed that treatment with rivaroxaban 5 mg bid, compared to acetylsalicylic acid (ASA), caused a significant increase in bleeding, in the absence of a clear clinical benefit. Instead, the rivaroxaban 2.5bid-ASA combination strategy proved to be more effective than ASA monotherapy, in terms of a 24% reduction in the combined primary endpoint (cardiovascular death, myocardial infarction, stroke). On the basis of these results, the recent guidelines of the European Society of Cardiology on chronic coronary syndromes recommend, in secondary prevention, the addition of a second antithrombotic drug to ASA in patients with high (recommendation class IIa, level of evidence A) or moderate (class of recommendation IIb, level of evidence A) risk of ischemic events, in the absence of high bleeding risk. The choice of drug to combine with ASA falls on a P2Y12 platelet receptor inhibitor or an anticoagulant, i.e. rivaroxaban 2.5 mg.

However, the use of the association of an antiplatelet drug with a low-dose anticoagulant drug and adherence to this treatment has not yet been adequately evaluated in the real world. In fact, no Italian observational data relating to this therapeutic strategy are currently available.

The observational, prospective, multicenter study includes patients suffering from symptomatic peripheral atherosclerotic disease of the lower limb, with or without chronic ischemic heart disease, and indication for treatment with rivaroxaban 2.5 mg bid and ASA 100 mg. The aim of the study is to examine the adherence to the treatment prescriptions after 3 months and after 12 months the enrolment and possible adverse events occurred in this time period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic peripheral atherosclerotic disease of the lower extremity
* Ability to provide written informed consent.

Exclusion Criteria:

* Need for dual antiplatelet therapy, or therapy with antiplatelet agents other than aspirin or oral anticoagulant therapy (full dose)
* Ischemic stroke within the previous 1 month or any history of hemorrhagic or lacunar stroke
* Dialysis or estimated glomerular filtration rate <15 mL/min
* Known non-cardiovascular disease associated with poor prognosis (e.g. metastatic cancer)
* History of known hypersensitivity to rivaroxaban, aspirin or excipients
* Presence of contraindications to rivaroxaban and/or aspirin (as indicated in the technical data sheet)
* Systemic treatment with strong inhibitors of CYP 3A4 or p-glycoprotein (e.g. systemic antifungals, such as ketoconazole and human immunodeficiency virus [HIV] protease inhibitors, such as ritonavir) or strong inducers of CYP 3A4, e.g. Rifampicin, Rifabutin, Phenobarbital, Phenytoin and Carbamazepine
* Any liver disease associated with coagulopathy
* Subjects who are pregnant, breastfeeding or potentially pregnant, or of childbearing age, sexually active and not practicing an effective method of birth prevention (e.g. prescription oral contraceptives, contraceptive injections, intrauterine device, double barrier method, patch contraceptive, sterilization of the male partner)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from symptomatic peripheral atherosclerotic disease of the lower limb, with or without chronic ischemic heart disease, and indication for treatment with rivaroxaban 2.5 mg bid and acetylsalicylic acid 100 mg
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to the prescribed medical treatment | 3 months
  Adherence to the prescribed medical treatment measured by the Morisky Medication. Adherence Scale. The scores range from 0 to 8, with scores of 8 reflecting high adherence, 7 or 6 reflecting medium adherence, and <6 reflecting low adherence.
Adherence to the prescribed medical treatment | 12 months
  Adherence to the prescribed medical treatment measured by the Morisky Medication Adherence Scale. The scores range from 0 to 8, with scores of 8 reflecting high adherence, 7 or 6 reflecting medium adherence, and <6 reflecting low adherence.

SECONDARY OUTCOMES:
Adverse event | 3 months
  Cardiovascular events, death
Adverse event | 12 months
  Cardiovascular events, death

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Scientifici Maugeri, Milan, Italy

IPD SHARING:
Plan to Share IPD: No